CLINICAL TRIAL: NCT05188690
Title: Clinical Presentation of COVID-19 Patients With an Associated Diagnosis of Polyneuropathy: a Multicenter Observational Study
Brief Title: Polyneuropathy and COVID-19
Acronym: PolyneuroCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Poliambulanza Istituto Ospedaliero (Other); Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor
Other Study IDs: FDG_multicenter_COVID19
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Polyneuropathies
Keywords: COVID-19; Polyneuropathy
MeSH Terms: conditions — COVID-19; Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection from medical records — Data collection from medical records

SUMMARY:
Since the onset of the Coronavirus pandemic disease 2019 (COVID-19), the Lombardy region and in particular the territory of the province of Brescia has been heavily affected. Current data show that the total number of confirmed cases in Italy of COVID-19 due to severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) exceeds 3.9 million cases, with more than 120 thousand deaths. As the COVID-19 epidemic continues to spread globally, more and more evidence is being gathered about the presence of neurological manifestations and symptoms associated with it. With the growing understanding of the disease, many non-pulmonary symptoms have been recognized, including neurological complications such as acute cerebrovascular disease, meningitis, encephalitis, and peripheral nervous system disease. The main objective of this study is to analyze the clinical and functional conditions of COVID-19 patients with an associated diagnosis of polyneuropathy who were admitted for rehabilitation in the rehabilitation centers of Brescia.

DETAILED DESCRIPTION:
The study will be conducted in all the centers considered following the same protocol based on data collection of COVID-19 patients with an associated diagnosis of polyneuropathy. Demographic information, clinical manifestations, laboratory results, electromyography (EMG), neuroimaging, and outcomes will be extracted from the medical records using a standardized data collection form. The data collection will be divided into demographic and clinical data, instrumental examinations, and functional assessment. In the section of demographic data will be collected information regarding age, sex, comorbidities (diabetes mellitus, dyslipidemia, hypertension, coronary artery disease, neoplasia, renal failure, anxiety-depressive syndrome or similar Etc. ), administration during hospitalization of antibiotics, antivirals, mechanical ventilation (invasive / non-invasive; Number of days of mechanical ventilation), pronation cycles (Yes / No), oxygen therapy (Yes / No; Number of days of oxygen therapy; L/min), time of hospitalization in an acute care facility (Number of days) and overall hospitalization time (Number of days). Concerning instrumental examinations will be collected data on neuroimaging tests (CT brain, MRI brain) and EMG more precisely: the type of polyneuropathy will be defined (axonal, demyelinating, mixed); the presence of conduction blocks (Yes/No); latency of F responses from posterior tibial; the amplitude of compound motor action potential (cMAP), distal latencies and motor conduction velocity of one nerve in the lower limbs and one in the upper limbs (possibly peroneal and ulnar); the presence of non-registrable responses (Yes/No); the amplitude of sural sensory-motor potential (SAP).

Data at admission and discharge will be collected on the: Cumulative Illness Rating Scale (CIRS), Barthel index, Modified Rankin scale (MRS), muscle strength of the four limbs (MRC muscle scale), walking (Autonomous, with aids, not autonomous). In terms of clinical outcomes will be considered the length of rehabilitation hospitalization (Number of days).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Sars-Cov2 infection, regardless of the degree of severity and negative results to 2 consecutive nasopharyngeal swabs.
* Diagnosis of Polyneuropathy is defined clinically and/or by electromyographic examination.
* Older age
* Both sexes

Exclusion Criteria:

* Presence of disabling conditions affecting the musculoskeletal system.
* Ischemic/hemorrhagic stroke
* Neurodegenerative diseases
* Presence of rheumatic and inflammatory diseases.
* Chronic diseases of the respiratory system.
* Hemodynamic instability
* Cognitive impairment (Mini-Mental State Examination <18)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of Sars-Cov2 infection, regardless of the degree of severity and negative results to 2 consecutive nasopharyngeal swabs. Diagnosis of Polyneuropathy is defined clinically and/or by electromyographic examination.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Barthel index | through study completion, an average of 6 months
  The Barthel Index (BI) is a measurement tool, based on an ordinal scale, commonly used to assess the Activities of Daily Living (ADLs) or all the basic activities that an adult individual performs independently and without the need for assistance to survive and take care of themselves.

SECONDARY OUTCOMES:
Cumulative Illness Rating scale (CIRS) | through study completion, an average of 6 months
  The Cumulative Illness Rating Scale is a reliable instrument for assessing physical impairment. Ratings are made on a 5-point "degree of severity" scale, ranging from "none" to "extremely severe."
muscle strength of the 4 limbs (MRC muscle scale). | through study completion, an average of 6 months
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Modified Rankin scale (MRs) | through study completion, an average of 6 months
  The Modified Rankin Scale (MR) is a scale for measuring the degree of disability in the daily activities.

OTHER OUTCOMES:
the length of rehabilitation hospitalization (Number of days) | through study completion, an average of 6 months
  Number of days in the rehabilitation center

CONTACTS AND LOCATIONS:
Locations (1):
- Centro "E. Spalenza - Don Gnocchi", Rovato, Italy

IPD SHARING:
Plan to Share IPD: Undecided